CLINICAL TRIAL: NCT03808324
Title: Allograft Vasculopathy and Unexplained Graft Dysfunction During Long-term Follow-up After Heart Transplantation
Brief Title: Heart Failure After Heart Transplantation Due to Chronic Rejection
Acronym: AVALON
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Sorosh Esmaily, Principal Investigator, Sahlgrenska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AVALON
Record Dates: First submitted 2018-12-29; First posted 2019-01-17 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Cardiac Allograft Vasculopathy; Chronic Rejection of Cardiac Transplant; Graft Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Heart transplant recipients (Experimental)
  Interventions: Diagnostic Test: Diagnostic investigations

INTERVENTIONS:
Diagnostic Test: Diagnostic investigations — Participants will undergo tests and diagnostics investigations to identify signs of chronic rejection after heart transplantation.

SUMMARY:
This study will investigate the prevalence of allograft vasculopathy and unexplained graft dysfunction during long-term follow-up after heart transplantation. Risk factors as well diagnostic approaches will be investigated.

DETAILED DESCRIPTION:
During long-term follow-up heart transplant recipients are at risk of developing different complications that are likely to affect quality of life and survival. The most common cause of death during the later stages after heart transplantation is cardiac allograft vasculopathy, followed by unexplained graft dysfunction. In this study, advanced imaging techniques will be used to describe the frequency of these two complications, examine possible risk factors and study consequences on functional capacity and quality of life. Further, the investigators will investigate whether it is feasible to screen for these conditions with non-invasive imaging methods. By studying patients that have performed cardiac transplantation between 10 and 20 years ago, the investigators expect to have a significant proportion of patients with these pathological conditions. Methods that will be used include cardiac magnetic resonance imaging, coronary flow velocity reserve assessment, right heart catheterization and coronary imaging with angiography and optical coherence tomography.

ELIGIBILITY:
Inclusion Criteria:

* Heart transplant performed more than 10 years and less than 21 years ago
* Scheduled yearly post-transplant control
* Signed informed consent

Exclusion Criteria:

* Estimated GFR < 30 mL/min/1,73m2
* Radiographic contrast allergy
* Severe asthma or COLD with FEV1 < 50%
* Second or third degree AV block
* Pregnancy
* In the Investigator's opinion, the patient has a clinically significant disease that could be adversely affected by study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Degree of stenosis in coronary arteries | 4 hours
  Coronary angiography gives information about the degree of stenosis in the coronary arteries. In connection with the angiography Optical Coherence Tomography (OCT) will be performed. A precise measurement and characterization of the intima can be performed by OCT.
Restrictive allograft hemodynamics | 2 hours
  Right heart catheterization will be performed using a Swan-Ganz pulmonary artery thermodilution catheter. Right atrial pressure (RAP), mean pulmonary artery pressure (MPAP), pulmonary capillary wedge pressure (PCWP) and mean arterial pressure (MAP). Cardiac output (CO) and cardiac index (CI) will be recorded by thermodilution. The transpulmonary gradient (TPG) is obtained by subtracting PCWP from MPAP and PVR (in Wood units (WU) by dividing TPG by CO. Measurement will be performed both at rest and after supine bicycle exercise. A restrictive allograft filling pattern will be defined as PCW at rest exceeding 15 mmHg and/or exceeding 25 mmHg during exercise.
Functional assessment of the microvasculature | 2 hours
  Coronary flow reserve (CRF) measurements may provide functional assessment of the microvasculature. Coronary blood flow velocity (CBFV) is measured in the left anterior descending coronary artery (LAD) before, and during constant adenosine infusion using conventional color Doppler ultrasound equipped with coronary imaging protocol. Mid-distal LAD segment is visualized using high frequency color Doppler (>3 MHz) in the anterior interventricular sulcus. A CINE-loop is then stored to document the 2-D image of LAD. Thereafter spectral Doppler is used to record CBFV. Mean diastolic flow velocity is calculated by manually tracing the diastolic flow velocity signal. Baseline CBFV values are calculated using the mean value of three representative heart beats during resting condition. The mean hyperemic CBFV is calculated as the mean of the three highest CBFV values recorded during the whole infusion period. The ratio between hyperemic and baseline CBFV is defined as CFR.
Degree of myocardial fibrosis | 4 hours
  Measurement of myocardial T1 times (T1 mapping) with gadolinium-enhanced inversion recovery-prepared sequences may depict diffuse myocardial fibrosis and has good correlation with ex vivo fibrosis content. T1 mapping calculates myocardial T1 relaxation times with image-based signal intensities and will be performed with standard cardiac MR imagers and radiologic workstations.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No